CLINICAL TRIAL: NCT00102726
Title: A Double-Blind, Randomized, Multicenter, Placebo-Controlled, Parallel Group, Dose Ranging Study to Assess the Efficacy, Safety, and Pharmacokinetics of an Oral Thrombopoietin Receptor Agonist(SB497115-GR) Administered at 50, 75, and 100 mg to Cancer Patients Receiving Multiple Cycles of Chemotherapy
Brief Title: SB-497115 (Oral Thrombopoietin Receptor Agonist) Versus Placebo In Adult Cancer Patients Receiving Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 497115/003
Record Dates: First submitted 2005-02-01; First posted 2005-02-02 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Thrombocytopaenia
Keywords: chemotherapy; thrombopoietin; platelets; chemotherapy induced
MeSH Terms: conditions — Thrombocytopenia; Jacobs syndrome | interventions — eltrombopag

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Arm 1 (Active Comparator): SB-497115-GR 50mg. administered orally daily on days 2 through 11 for each 21-day cycle.
  Interventions: Drug: SB497115
- Arm 2 (Active Comparator): SB-497115-GR 75 mg administered orally dailey on days 2-11 of each 21-day cycle.
  Interventions: Drug: SB497115
- Arm 3 (Active Comparator): SB-497115 100mg administered orally daily on days 2 through 11 of each 21-day cycle.
  Interventions: Drug: SB497115
- Placebo Arm (Placebo Comparator): Placebo administered orally daily on days 2 through 11 of each 21-day cycle.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: SB497115 — SB497115/Placebo will be administered for at least 2 cycles. Additional cycles are permited if: 1) chemotherapy is continued, 2) the subject appears to be benefitting from the study drug, and 3) the subject has not encountered greater than moderate toxicity with the study drug. The maximum number of cycles would be 8.
  Arms: Arm 1; Arm 2; Arm 3
Other: Placebo — Placebo administered orally daily on days 2 through 11 of each 21-day cycle.
  Arms: Placebo Arm

SUMMARY:
SB497115 is an oral agent which activates the thrombopoietin receptor and increases platelet counts in healthy volunteers. This study is examining several different doses of SB497115 versus placebo as treatment for patients with advanced solid tumors scheduled to receive chemotherapy with carboplatin and paclitaxel every 21 days. Patients will receive SB497115 on days 2-11 of each 21 day cycle for at least 2 cycles of chemotherapy and for a maximum of 8 cycles of chemotherapy.

DETAILED DESCRIPTION:
A Double-Blind, Randomized, Multicenter, Placebo-Controlled, Parallel Group, Dose Ranging Study to Assess the Efficacy, Safety, and Pharmacokinetics of an Oral Thrombopoietin Receptor Agonist (SB-497115-GR) Administered at 50, 75, and 100 mg to Cancer Patients Receiving Multiple Cycles of Chemotherapy

ELIGIBILITY:
Inclusion criteria:

* Subjects ≥18 years old, who are chemotherapy naïve, with histologically or cytologically confirmed advanced solid tumor (leukemia and lymphoma are excluded) who are scheduled to received carboplatin/paclitaxel as shown below. For the purpose of this study, advanced tumors are defined as tumors that are being treated with palliative intent (i.e., not being treated with curative intent).
* Subjects scheduled to receive first-line chemotherapy as carboplatin AUC 5-6 IV over 30 minutes plus paclitaxel 175-225 mg/m2 IV over 3 hours on day 1 every 21 days, with routine pre-medications, i.e., 20 mg dexamethasone [or equivalent] orally 6 and 12 hours pre-paclitaxel, 50 mg IV diphenhydramine [or equivalent] and 300 mg IV cimetidine [or equivalent] 30-60 minutes pre-paclitaxel.
* ECOG-Zubrod performance status is 0, or 1.
* Subject has no history of platelet disorders or dysfunction and no history of a bleeding disorder.
* Subjects have adequate:

hematologic function (ANC ≥ 1,500/mm3, hemoglobin ≥ 9 g/dL, and platelet count ≥100,000/mm3 and < upper limit of normal range (eg, 400,000 to 450,000/mm3), hepatic function (bilirubin ≤ 2 mg/dL and alanine aminotransferase ≤ three times the upper limit of normal), renal function (creatinine ≤ 2.0 mg/dL).

* Subject has no physical limitation to ingest and retain oral medication.
* Subject has life expectancy of at least 6 months.
* Subject is practicing an acceptable method of contraception (documented in chart). Female subjects (or female partners of male subjects) must either be of nonchildbearing potential (hysterectomy, bilateral oophorectomy, bilateral tubal ligation or post-menopausal > 1 year), or of childbearing potential and use one of the following acceptable methods of contraception from two weeks prior to administration of study medication, throughout the study, and 28 days after completion or premature discontinuation from the study:

Complete abstinence from intercourse; Intrauterine device (IUD); Two forms of barrier contraception (diaphragm plus spermicide, and for males condom plus spermicide); Male partner is sterile prior to entry into the study and is the only partner of the female; Systemic contraceptives (combined or progesterone only).

* Subject is able to understand and comply with protocol requirements and instructions and intend to complete the study as planned.
* Subject has signed and dated written informed consent.
* Chemotherapy naive patients with advanced solid tumors (without brain metastasis or rapid progression within 2 weeks) who are scheduled to receive standard first-line therapy with carboplatin and paclitaxel every 21 days.
* Adequate hematologic, hepatic and renal function.

Exclusion criteria:

* Any clinically relevant abnormality, other than cancer, identified on the screening examination, or any other medical condition or circumstance, which in the opinion of the Investigator, makes the subject unsuitable for participation in the study and/or would make the patient's data difficult to interpret.
* Subjects with a known history of rapidly progressive disease (marked increase in tumor size [>50%], ascites, or serious symptoms related to underlying cancer in the preceding 4-week period), surgery within the previous 2 weeks, radiotherapy within the previous 4 weeks, or any prior chemotherapy.
* Subjects with known pre-existing cardiac disease, including congestive heart failure, arrhythmias requiring treatment, or myocardial infarction within the preceding 3 months.
* Subjects with abnormal resting 12-lead ECG at screening that would indicate preexisting cardiac disease, as noted in exclusion criterion 3.
* Subjects with known clotting disorder associated with hypercoaguability.
* Subject has consumed aspirin, aspirin-containing compounds, salicylates, quinine or non-steroidal anti-inflammatories (NSAIDs) for > 3 consecutive days within 2 weeks of the study start and would require them at any time during the study.
* Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of study medication.
* Subject has consumed liquid antacids (e.g. Maalox, Mylanta, Amphogel, milk of magnesia), chewable antacids (e.g. TUMS) or calcium supplements within 48 hours of the first dose of study medication, and/or will require these medications during the study.
* Subject has consumed rosuvastatin or pravastatin within 1 week of the first dose of study medication and/or will require these medications at any time during the study.
* Any history of drug-induced thrombocytopenia (e.g., quinine).
* Systemic anti-coagulant use within 4 weeks prior to study entry.
* Consumption of any herbal or dietary supplements, excluding vitamin or mineral supplements (See Exclusion 8 for calcium supplements), within 1 week of the study start.
* Female subjects who are lactating or have a positive beta-hCG at screening.
* Subjects with a history of CNS metastases or clinical signs or symptoms of brain and/or leptomeningeal metastases confirmed by CT or MRI brain scan.
* History of platelet or bleeding disorders.
* Patients using aspirin, aspirin-containing compounds, salicylates, antacids, rosuvastatin, pravastatin, non-steroidal anti-inflammatory drugs for greater than 3 days during and within 3 weeks prior to the study.
* Females who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2005-02; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Change in baseline platelet count from the first day of the second cycle of chemotherapy to the lowest count observed (nadir) during the cycle(21 days) | throughout entire study

SECONDARY OUTCOMES:
Safety and tolerability, pharmacodynamics, changes in platelet count during cycle 1(21 days) and beyond cycle 2(21 days), population PK, and deliver intended doses of chemotherapy without thrombocytopenia related AEs | Throughout entire study
Safety and tolerability as indicated by physical exam, 12-lead ECGs, ophthalmologic examinations, clinical laboratory tests, clinical monitoring/observation, and AE reporting | throughout study
Pharmacodynamic parameters including platelet count, grade of thrombocytopenia,serum thrombopoietin, and platelet aggregation/activation during the first and second cycles of carboplatin/paclitaxel | During first and second cycles of carboplatin/paclitaxel
Change in platelet count from day 1 (baseline) to nadir during the first cycle and beyond the second cycle of carboplatin/paclitaxel | throughout study
Population PK of SB-497115, including clearance (CL/F), absorption rate constant(ka), and volume of distribution (V/F) with assessment of demographic covariates influencing SB-497115 PK | throughout study
The relationship between PK of SB-497115 andrelevant safety and efficacy endpoints will be explored | throughout study
Dose intensity (percent of intended dose) of carboplatin/paclitaxel
Carboplatin/paclitaxel-associated thrombocytopenia-related AEs, as defined by NCI
Common Terminology Criteria for Adverse Events, CTCAE v3.0, to include the number of platelet transfusions, bleeding events (hematoma), hemorrhage/bleeding,petechiae/purpura), clinical laboratory tests, and clinical observations | throughout study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (84):
- United States (26):
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Greenbrae, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Newark, Delaware
  - GSK Investigational Site, Boca Raton, Florida
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Tamarac, Florida
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Hattiesburg, Mississippi
  - GSK Investigational Site, Tupelo, Mississippi
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Babylon, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Mayfield Heights, Ohio
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Bryan, Texas
  - GSK Investigational Site, Ogden, Utah
  - GSK Investigational Site, Salem, Virginia
- Argentina (5):
  - GSK Investigational Site, Buenos Aires, Buenos Aires
  - GSK Investigational Site, Capital Federal, Buenos Aires
  - GSK Investigational Site, La Plata, Buenos Aires
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Buenos Aires
- GSK Investigational Site, Vienna, Austria
- Bulgaria (2):
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Sofia
- Czechia (2):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Prague
- Germany (9):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Regensburg, Bavaria
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Marburg, Hesse
  - GSK Investigational Site, Hemer, North Rhine-Westphalia
  - GSK Investigational Site, Trier, Rhineland-Palatinate
  - GSK Investigational Site, Großhansdorf, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin
  - GSK Investigational Site, Bad Berka, Thuringia
- Hungary (2):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Székesfehérvár
- India (4):
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Hyderabad, Andhra Pradesh
  - GSK Investigational Site, Kolkata
  - GSK Investigational Site, Vellore
- Italy (4):
  - GSK Investigational Site, Benevento, Campania
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Campobasso, Molise
- GSK Investigational Site, Mérida, Yucatán, Mexico
- GSK Investigational Site, Lima, Lima Province, Peru
- Poland (4):
  - GSK Investigational Site, Olsztyn
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Szczecin
  - GSK Investigational Site, Wroclaw
- GSK Investigational Site, Bucharest, Romania
- Russia (3):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Moscow Region
  - GSK Investigational Site, Saint Petersburg
- GSK Investigational Site, Seoul, South Korea
- Spain (7):
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Santa Cruz de Tenerife
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Seville
- Taiwan (2):
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Tau-Yuan County
- Ukraine (4):
  - GSK Investigational Site, Dnipro
  - GSK Investigational Site, Donetsk
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Lviv
- United Kingdom (5):
  - GSK Investigational Site, Truro, Cornwall
  - GSK Investigational Site, Chelmsford, Essex
  - GSK Investigational Site, Colchester
  - GSK Investigational Site, Dundee
  - GSK Investigational Site, Leicester

REFERENCES:
- [Background] Hayes S, Mudd PN Jr, Ouellet D, Johnson BM, Williams D, Gibiansky E. Population PK/PD modeling of eltrombopag in subjects with advanced solid tumors with chemotherapy-induced thrombocytopenia. Cancer Chemother Pharmacol. 2013 Jun;71(6):1507-20. doi: 10.1007/s00280-013-2150-9. Epub 2013 Apr 6. PMID 23564375
- [Background] Kellum A, Jagiello-Gruszfeld A, Bondarenko IN, Patwardhan R, Messam C, Mostafa Kamel Y. A randomized, double-blind, placebo-controlled, dose ranging study to assess the efficacy and safety of eltrombopag in patients receiving carboplatin/paclitaxel for advanced solid tumors. Curr Med Res Opin. 2010 Oct;26(10):2339-46. doi: 10.1185/03007995.2010.510051. PMID 20735290